CLINICAL TRIAL: NCT06963385
Title: Correlation Between RadiOmics and Molecular Classification in Endometrial Cancer (the ROME Study): a Step Forward to a Simplified Precision Medicine
Brief Title: Radiomics and Molecular Classification in Endometrial Cancer
Acronym: ROME
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Principal Investigator, Valentina Chiappa, M.D., Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Int140/20
Record Dates: First submitted 2020-12-01; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Endometrial Cancer; Uterine Cancer; Endometrium Tumor
Keywords: radiomics; endometrial cancer; molecular/genetic profiling; radiogenomics; ultrasound
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Neoplasms | interventions — Radiomics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radiomics analysis and molecular/genomic profiling (Experimental): This prospective single-arm observational study. Patients with newly diagnosed endometrial cancer have an ultrasonographic evaluation and radiomic analysis of the ultrasonographic images. Then patients have surgery followed by molecular/genomic evaluation. We correlate radiomic features with molecular/genomic profiling.
  Interventions: Diagnostic Test: Radiomics

INTERVENTIONS:
Diagnostic Test: Radiomics — To correlate radiomic features obtained from ultrasound images with the molecular/genomic profiling to identify new hallmarks for stratification of endometrial cancer patients into different classes of risk

SUMMARY:
Molecular/genomic profiling is the most accurate method to assess the prognosis of endometrial cancer patients. Interestingly, the adoption of radiomics showed important results, across various oncologic specialties. Radiomic allows extracting mineable high-dimensional data from clinical images, thus providing a number of noteworthy information of the tumor tissues. We aim to correlate radiomic features obtained from ultrasound images with the molecular/genomic profiling to identify new hallmarks for stratification of endometrial cancer patients into different classes of risk The central hypothesis is that combining radiomic features might allow identifying various classes of risk for endometrial cancer. The rationale for the proposed research is that once validated, radiomics applied to ultrasonographic images would be an effective, innovative, and cheap method for tailor operative and postoperative treatment modality in endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

(i) preoperative endometrial cancer (any histology); (ii) preoperative ultrasonographic examination; (iii) surgical treatment; (iv) age >= 18 years; (v) signed informed consent for research purposes.

Exclusion Criteria:

(i) consent withdraw; (ii) lack of available (tumor) tissue for molecular/genomic profiling.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients affected by endometrial cancer
Enrollment: 250 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To detail the mechanism by which radiomic features predict the classification of endometrial cancer into various classes of risk. | 1-18 months
Determinate the scaled impact of radiomic features assessed on ultrasonographic images of endometrial tumors. | 1-36 months

SECONDARY OUTCOMES:
Assess the intraobserver and interobserver reproducibility of radiomic features on ultrasonographic images of endometrial tumors | 19-36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori di Milano, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided